CLINICAL TRIAL: NCT05090072
Title: Advanced Directives in Palliative Care: Physician's Role on Caregiver's Empowerment as Patient's Surrogates
Brief Title: Advanced Directives in Palliative Care (DAVPAL)
Acronym: DAVPAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Catarina Sampaio Martins, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DAVPAL Study
Record Dates: First submitted 2021-09-28; First posted 2021-10-22 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: End-of-life
Keywords: palliative care; Advance Directives; caregivers; End-of-life decision-making
MeSH Terms: conditions — Death | interventions — Advance Directives

STUDY DESIGN:
Intervention Model Description: After enrollment and some sociodemographic data were collected, participants were asked to, separately, fulfill the Advance Directives document, concerning patients' last wishes. Caregivers also fulfill one document with their own end-of-life preferences.
  The pair was then randomly assigned to one of the two parallel groups (Advance Directives or Control Group).
  Both groups had a conference meeting with the same palliative care physician, in the same room, with the same average duration (40 to 50 minutes). The Advance Directives Group discussed patients' answers to the Advance Directive document, and the Control Group talked about patients' clinical status.
  Two months later, caregivers only, were asked to fulfill another Advance Directive document as patients' surrogates.
Who Masked: Participant
Masking Description: All participants were blinded to the allocated intervention, from the beginning to the end of the trial. Investigator only had access to the allocation group after participants enrollment on the trial, sociodemographic data collected, and phase 1 Advance Directives fulfilled.
  Preliminary data analysis was made without knowledge of the participants' allocated group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- - Advance Directives Group (Active Comparator): The group that will receive the principal physician intervention, using Advance Directives document as a communication tool between patients and caregivers, to find its efficacy on the promotion of better-prepared surrogates
  Interventions: Behavioral: Advance Directives
- Control Group (Placebo Comparator): The group that will receive the Placebo Intervention, consisting of a clinical evaluation of patients' clinical status, by the physician
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Advance Directives — The palliative care physician engaged patients and their caregivers in an open discussion about patients' answers to the Advance Directives document, to explore and clarify all doubts and questions prompted by the document
  Arms: - Advance Directives Group
Behavioral: Control — The palliative care physician undergone a conference with both patients and caregivers and evaluated patients' symptoms using the the Edmonton Frail Scale (Bruera, 1991), adapted to the Portuguese population. The Advance Directives theme wasn't approached during this conference.
  Arms: Control Group

SUMMARY:
A prospective, single-blinded, controlled, and randomized trial to find if physician's use of the Portuguese Advance Directives, in palliative care, as a communication tool between patients and caregivers, improves the agreement and reliability between patients and their health surrogates, in their decisions about end-of-life care.

DETAILED DESCRIPTION:
This trial was a prospective, single-blinded, controlled, and randomized study analyzing if Advance Directives' discussion between patients and caregivers, promoted by a palliative care physician, improves concordance between them, concerning to patients' last wishes, therefore improving surrogates' accuracy when caregivers decide and act on behalf of the patients. This trial was conducted in a central hospital of Portugal's north inland, serving an estimated population of 465.000 habitants. Patients referenced to all three units of the palliative care service from September 2018 to September 2019, and caregivers, were sequentially approached and recruited on the first consult.

All participants gave written consent to enroll in the trial. This study occurred in two phases, within a 1-month interval. At baseline (phase 1) participants separately fulfilled the Advance Directives' document considering patients' preferences for end-of-life care. Caregivers also fulfill a similar document with their own end-of-life preferences.

Dyads were then randomly assigned to two different groups - The Advance Directives and the Control groups.

Simple individual randomization was previously informatically achieved and the randomization sequence was disclosed by a sealed envelope only after trial enrollment of the dyad, to ensure proper investigator concealment. Both patients and caregivers were blinded to the assigned group until the end of the trial. In both groups (Advance Directives and Control), dyads were engaged in a conference meeting, in the same room, with the same average duration, with the same investigator.

In the Advance Directives group, the palliative care physician promoted an open discussion between patients and caregivers, about patients' answers to the Advance Directives document. In the Control group, the palliative care physician underwent a conference with both patients and caregivers to evaluate patients' clinical symptoms.

At phase 2, one month after the first interview, caregivers were asked to fill in another Advance Directives document, as patients´ surrogates.

Each participant had the choice to drop out at any moment of the trial, and the pair was excluded from data analysis.

Portuguese official Advance Directives was the central instrument used in this trial. Participants were asked to choose 1 to 3 different scenarios, to apply the following 12 questions regarding end-of-life preferences. Each question in each scenario was informatically registered as a Yes or No item, respectively corresponding to items selected or not by all participants. For each participant, the investigators expected 36 possible answers for concordance analysis.

Categorical variables were described by absolute and relative frequencies. Age was described by the mean and standard deviation (mean ± SD), as its distribution was not deviated from normality in each group, according to visual analysis of histograms and confirmed with the Shapiro-Wilk's test of normality.

Agreement between patients and caregivers was assessed (in each question) with the Overall Proportions of Agreement (Overall PA) and Proportions of Specific Agreement (for Yes and No), with respective 95% confidence intervals. Reliability was accessed with Cohen's kappa (k).

Descriptive data analysis was performed using SPSS® Statistics. Proportions of agreement and Cohen's κ with respective confidence intervals were computed using packages "obs. agree" and "psych" from R software, v 3.4.0.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with 18 years or more
* Patients referenced to the palliative care service with a chronic, progressive, and incurable disease
* Patients with the ability to comprehend, write and speak the Portuguese language
* Patients with an absence of major cognitive disorders (Portuguese validated Mini-Mental State Test score superior to 22, 25, or 27, according to patients' scholarly)
* Patients that accepted to participate in the trial
* Patients who were capable of nominate a caregiver as their surrogate in decision making
* Adult caregivers with 18 years or more
* Caregivers who were nominated by patients as their surrogate decision-maker
* Caregivers with the ability to comprehend, write and speak the Portuguese language
* Caregivers that accepted to participate in the trial

Exclusion Criteria:

* Patients or caregivers that refused to participate
* Patients with cognitive impairment
* Patients with incapacity to dialogue
* Patients who were too sick to cooperate
* Patients without a caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Agreement between patients´ and caregivers´ answers in the Advance Directives´ document | 1 month
  Agreement between patients and their caregivers was accessed with the Overall Proportion of Agreement (Overall PA) and Proportion of Specific Agreement (Yes PA and No PA), for the 12 questions of the Portuguese Advance Directives, on the Advance Directives and Control group
Reliability of the results of agreement between patients´ and caregivers' answers in the Advance Directives´ document | 1 month
  Reliability was accessed with Cohen's kappa (k). (Cohen, 1960). We assumed Landis and Koch's (1977) interpretation of κ value. According to these authors, a κ value of 0.20 represents slight reliability, a value between 0.21 and 0.40 fair reliability, a value between 0.41 and 0.60 moderate reliability, a value between 0.61 and 0.80 substantial reliability, and a value of 0.81-1.00 indicates almost perfect reliability

SECONDARY OUTCOMES:
Agreement between caregivers' answers as patients' surrogates and caregivers' answers about their own end-of-life preferences | 1 month
  Agreement between caregivers as surrogates and their own preferences was accessed with the Overall Proportion of Agreement (Overall PA) and Proportion of Specific Agreement (Yes PA and No PA), for the 12 questions of the Portuguese Advance Directives, on the Advance Directives and Control group

CONTACTS AND LOCATIONS:
Locations (1):
- Tràs-os-Montes and Alto Douro Hospital Centre, Vila Real, Portugal

REFERENCES:
- [Derived] Martins CS, Nunes R. Portuguese Advance Directives-a twist against futility? A cross sectional study. Sao Paulo Med J. 2024 Mar 25;142(3):e2022537. doi: 10.1590/1516-3180.2022.0537.R2.201023. eCollection 2024. PMID 38536997
- [Derived] Martins CS, Nunes R. Advanced directives' knowledge among Portuguese palliative patients and caregivers: do the sociodemographic factors influence it? A cross-sectional survey. BMC Palliat Care. 2023 Jul 1;22(1):84. doi: 10.1186/s12904-023-01203-7. PMID 37393243
- [Derived] Martins CS, Sousa I, Barros C, Pires A, Castro L, da Costa Santos C, Nunes R. Do surrogates predict patient preferences more accurately after a physician-led discussion about advance directives? A randomized controlled trial. BMC Palliat Care. 2022 Jul 12;21(1):122. doi: 10.1186/s12904-022-01013-3. PMID 35820845

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT05090072/Prot_SAP_000.pdf
  • Informed Consent Form: Patient Informed Consent (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT05090072/ICF_001.pdf
  • Informed Consent Form: Caregiver Informed Consent (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT05090072/ICF_002.pdf